CLINICAL TRIAL: NCT06794502
Title: Interferon Gamma, Interleukin-10, Hematology and Microscopic Profile of Tuberculosis Patients With Treatment Combination of Anti-Tuberculosis and Butterfly Pea Flowers Extract (Clitoria Ternatea)
Brief Title: Butterfly Pea Flower (Clitoria Ternatea) for Adjuvant TB Treatment
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Universitas Muhammadiyah Semarang (Other)
Responsible Party: Principal Investigator, Maya Dian Rakhmawatie, Dr. MSc., Universitas Muhammadiyah Semarang
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UMuhammadiyahSemarang; 108/E5/PG.02.00.PL/2024 (Other Grant/Funding Number: Ministry of Research, Technology, and Higher Education of the Republic of Indonesia)
Record Dates: First submitted 2025-01-20; First posted 2025-01-27 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Tuberculosis (TB); Tuberculosis Treatment Effectiveness
Keywords: Anti-inflammatory agents; Butterfly pea flower; Cytokines; Tuberculosis therapy; Clitoria ternatea
MeSH Terms: conditions — Tuberculosis | interventions — Phytotherapy; Therapeutics

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Butterfly pea flower extract and anti-TB regimens (Active Comparator): The adjuvant therapy group of Tuberculosis patients (Group 1) were given an herbal medicine butterfly pea flower extract of 40 mL/day and anti-TB regimen for 2 months.
  Interventions: Drug: Herbal medicine
- Anti-TB regimens monotherapy (Other): The patients in anti-TB monotherapy group (Group 2) were given a regimen consisting of rifampicin, isoniazid, pyrazinamide, and ethambutol for 2 months.
  Interventions: Other: Tuberculosis (TB) treatment

INTERVENTIONS:
Drug: Herbal medicine — Herbal medicine from butterfly pea flower decocta extract is used as an additional TB drug therapy regimen for active TB patients during the initiation phase of treatment for 2 months.
  Other Names: Decocta extract of Clitoria ternatea; Butterfly pea flower extract
  Arms: Butterfly pea flower extract and anti-TB regimens
Other: Tuberculosis (TB) treatment — The patients in anti-TB monotherapy group (Group 2) were given a regimen consisting of rifampicin, isoniazid, pyrazinamide, and ethambutol for 2 months. This group did not receive any additional therapy.
  Arms: Anti-TB regimens monotherapy

SUMMARY:
The goal of this clinical trial is to learn if butterfly pea flowers (Clitoria ternatea) decocta extract works to treat as adjuvant therapy for tuberculosis in adults. It will also learn about the safety of butterfly pea flowers decocta extract.

The main questions it aims to answer are:

* Does butterfly pea flower extract as an adjunct TB drug therapy drug affect the profiles of interferon gamma and interleukin-10 of people with tuberculosis?
* Does butterfly pea flower extract as an adjunct TB drug therapy drug affect the hematology profiles of people with tuberculosis?
* Does butterfly pea flower extract as an adjunct TB drug therapy drug affect the clinical symptoms and acid-fast bacilli microscopic analysis of people with tuberculosis?
* What medical problems do participants have when taking butterfly pea flower decocta extracts?

Researchers will compare butterfly pea flower extract as an adjunct TB drug therapy to monotherapy TB drugs to see if adjuvant butterfly pea flowers extract works to treat tuberculosis infection in 2-month initiation phase therapy.

Participants will:

* Take drug butterfly pea flower extract plus TB regimen drugs consisting of rifampicin, isoniazid, pyrazinamide, and ethambutol or monotherapy TB regimen drugs only every day for 2 months
* Willing to undergo treatment monitoring and visit the clinic once every 2 weeks for checkups and tests
* Keep a diary of their symptoms and the number of times they use a butterfly pea flower decocta extract

ELIGIBILITY:
Inclusion Criteria:

* Pulmonary TB patients were positive based on the results of the Rapid Molecular Test GeneXpert M. tuberculosis (MTB)/Rifampicin (RIF),
* Patients who were undergoing the initiation phase of anti-TB treatment for the first time,
* Non-Multi Drug Resistant (MDR)/Extensively-Drug Resistant (XDR) TB patients with first-line anti-TB treatment (rifampicin, isoniazid, pyrazinamide, and ethambutol),
* Patients >18 years old,
* Patients who were willing to become research subjects and signed informed consent.

Exclusion Criteria:

* TB patients with Human Immunodeficiency Virus (HIV) positive,
* Patients who did not complete the study,
* Patients with non-compliance in taking medication,
* Patients with comorbidities (autoimmune and cancer),
* Smoking patients,
* Patients contraindicated in using butterfly pea flower extract.

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2024-03-14 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
The interferon-gamma and interleukin-10 cytokines | From enrollment to the end of treatment at 2 months
  Evaluation of the success of anti-TB therapy and anti-TB plus adjuvant butterfly pea flower therapy was carried out after completion of the 2-month initiation phase of treatment. Change Factor Analysis (CFA) for each cytokines parameter (interferon gamma or interleukin 10) was compared between the two treatment groups. Change Factor Analysis (CFA) for each therapy group was used to see whether there was an increase or decrease in cytokine concentrations after 2 months of therapy. The value was calculated from the concentration of each cytokine after treatment minus the concentration before treatment and divided by the concentration before treatment. After obtaining the CFA value for each group, the results between the groups were compared using independent t-test analysis.
Hematology profiles | From enrollment to the end of treatment at 2 months
  For hematological profile analysis, the Change Factor Analysis (CFA) for each parameter, namely Hb (g/dL), leukocytes and platelets (cells/µL), hematocrit and granulocytes (%), and Erythrocyte Sedimentation Rate (ESR) (mm/hour) was calculated for each treatment group. Change Factor Analysis (CFA) in each therapy group was used to see whether there was an increase or decrease in the concentration of each hematological parameter after 2 months of therapy. This CFA value is calculated from the concentration of each hematological profile after treatment minus the concentration before treatment and divided by the concentration before treatment. After obtaining the CFA value for each hematology parameter in each group, the results between butterfly pea flower extract plus anti TB-regimen groups and monotherapy anti-TB regimen were compared using independent t test analysis.
Microscopic profiles of acid-fast bacilli (AFBs) | From enrollment to the end of treatment at 2 months
  Microscopic analysis of Mycobacterium tuberculosis was carried out using Ziehl-Nielsen staining of sputum from TB patients in all therapy groups. Microscopic examination was carried out before and after treatment. The results of the examination are evaluated descriptively by seeing whether there is a decrease in the positive value of the number of colonies found during the examination.

OTHER OUTCOMES:
Clinical symptoms and toxicity | From enrollment to the end of treatment at 2 months
  Evaluation of clinical symptoms is carried out before and after therapy, by looking at whether there is an improvement in the symptoms of fever, cough, shortness of breath in TB patients. Hepatic toxicity was evaluated by observing whether jaundice occurred or not.

CONTACTS AND LOCATIONS:
Overall Officials: Sri Darmawati, Professor, Principal Investigator — Universitas Muhammadiyah Semarang
Locations (2):
- Indonesia (2):
  - West Kotawaringin Health Department, Pangkalanbuun, Central Kalimantan
  - Mendawai Community Health Center, Pangkalanbuun, Central Kalimantan